CLINICAL TRIAL: NCT02568098
Title: Open-Label Study to Evaluate Safety, Tolerability, Potential Pharmacokinetic Interactions and Mosquito-Lethal Effects of Orally Administered Ivermectin, Primaquine, Dihydroartemisinin-Piperaquine, and Albendazole in Healthy Adult Subjects
Brief Title: Pharmacokinetic and Mosquito-Lethal Effects of Ivermectin (IVM), Primaquine (PQ), Dihydroartemisinin-Piperaquine (DHA-PQP) and Albendazole (ABZ) in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Mahidol University (Other); Mahidol Oxford Tropical Medicine Research Unit (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FTM1501
Record Dates: First submitted 2015-05-26; First posted 2015-10-05 (Estimated); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Drug Combination; Pharmacokinetics; Healthy
Keywords: Drug combination; Ivermectin; Primaquine; Dihydroartemisinin-Piperaquine; Albendazole; Pharmacokinetics; Mosquito-Lethal Effect; Healthy adult subject
MeSH Terms: interventions — Intravital Microscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- TMEC-14-022 (OxTREC 39-14) (Experimental): Subjects had previously taken drug CQ and PQ
  Interventions: Drug: IVM, IVM and PQ, IVM and DHA-PQP, IVM and DHA-PQP and PQ; Drug: PQ and DHA-PQP and PQ
- TMEC 12-004 (OxTREC 58-11) (Experimental): Subjects had previously taken drug PQ and DHA-PQP
  Interventions: Drug: IVM, IVM and PQ, IVM and DHA-PQP, IVM and DHA-PQP and PQ
- New subject (Experimental): Subjects who not previously participated in study "TMEC 12-004 (OxTREC ref. 58-11)" and study "TMEC 14-022 (OxTREC ref. 39-14)".
  Interventions: Drug: IVM, IVM and PQ, IVM and DHA-PQP, IVM and DHA-PQP and PQ; Drug: PQ and DHA-PQP and PQ; Drug: DHA-PQP

INTERVENTIONS:
Drug: IVM, IVM and PQ, IVM and DHA-PQP, IVM and DHA-PQP and PQ — Regimen 1: IVM; Regimen 2: IVM and PQ; Regimen 3: IVM and DHA-PQP; Regimen 4: IVM and DHA-PQP and PQ;
Drug: PQ and DHA-PQP and PQ — Regimen 5: PQ; Regimen 7: DHA-PQP and PQ
  Arms: New subject; TMEC-14-022 (OxTREC 39-14)
Drug: DHA-PQP — Regimen 6: DHA-PQP
  Arms: New subject

SUMMARY:
Primary Objective

* To evaluate the safety and tolerability of co-administered single dose Dihydroartemisinin-Piperaquine (DHA-PQP), Ivermectin (IVM), Primaquine (PQ), and Albendazole (ABZ) in healthy subjects.

Secondary Objectives

* To characterize the potential pharmacokinetic interactions between DHA-PQP, IVM, PQ, and ABZ in healthy adult subjects.
* To characterize the pharmacokinetic properties of PQ (and its major metabolite), DHA-PQP, IVM, and ABZ (and its major metabolite) when given alone and in combination.
* To investigate pharmacogenetic polymorphisms affecting drug levels of PQ, DHA-PQP, IVM, ABZ and their metabolites.
* To determine mosquito lethal efficacy of IVM, PQ, ABZ, and DHA-PQP combinations against Anopheles dirus and Anopheles minimus.
* To determine if IVM concentrations in venous blood differs from capillary blood.

DETAILED DESCRIPTION:
This is an open-label, sequential pharmacokinetic study in 16 healthy glucose-6-phosphate dehydrogenase (G6PD) normal Thai subjects. These 16 subjects have previously participated in either study:

1. Open-Label Study to Evaluate Potential Pharmacokinetic Interaction of Orally Administered Primaquine (PQ) and Dihydroartemisinin-Piperaquine (DHA-PQP) in Healthy Adult Subjects (TMEC 12-004 (OxTREC ref. 58-11)) or study
2. Comparison of the electrocardiographic effects in relation to Pharmacokinetic profile of chloroquine (CQ) and piperaquine (PQ) in healthy Thai subjects (TMEC 14-022 (OxTREC ref. 39-14)) or
3. subjects who not previously participated in study "TMEC 12-004 (OxTREC ref. 58-11)" and study "TMEC 14-022 (OxTREC ref. 39-14)".

The study team will use the results of DHA-PQP regimen of the subjects from the above mentioned studies to compare with combination regimens in this study. This is to avoid unnecessary exposure of Subjects from (TMEC 12-004 (OxTREC ref. 58-11)) and (TMEC 14-022 (OxTREC ref. 39-14)) to the subjects. In addition, subjects have previously been tested for G6PD deficiency during screening process from the above mentioned study with result showed as normal. Therefore, a G6PD deficiency test is not needed. A G6PD deficiency test is needed for subjects who not previously participated in study subjects who not previously participated in study "TMEC 12-004 (OxTREC ref. 58-11)" and study "TMEC 14-022 (OxTREC ref. 39-14)" for this study.

Subjects will be admitted in the inpatient ward to receive single dose of 6 regimens (regimens 1-4 and 8-9) described below. Every subject will have at least 6 admissions in the hospital.

1: IVM (400 μg/kg) via 6 mg tabs, w-o** >4wks; 2: IVM (400 μg/kg)+PQ (15 mg): 2 tabs), w-o >4wks; 3: IVM (400 μg/kg)+DHA-PQP (40mg/320 mg): 3 tabs), w-o >8wks; 4: IVM (400 μg/kg)+DHA-PQP+PQ, w-o >8wks; 5*#: PQ (15 mg): 2 tabs, w-o > 2wks; 6#: DHA-PQP (40mg/320 mg): 3 tabs, w-o >8wks; 7*#: DHA-PQP (40mg/320 mg): 3 tabs +PQ (15 mg): 2 tabs, w-o >8wks; 8: ABZ (200 mg) 2 tabs, w-o >2wks; 9: IVM (400 μg/kg)+DHA-PQP (40mg/320 mg): 3 tabs+PQ (15 mg): 2 tabs +ABZ (400 mg): 1 tab, w-o >8wks

* The subjects from TMEC-14-022 (OxTREC ref. 39-14) will have two additional admissions to receive two additional regimen PQ, and DHA-PQP with PQ

# Subjects who not previously participated in study "TMEC 12-004 (OxTREC ref. 58-11)" and study "TMEC 14-022 (OxTREC ref. 39-14)" will have three additional admissions to receive three additional regimens PQ, DHA-PQP, and DHA-PQP with PQ.

**w-o = washout period

ELIGIBILITY:
Inclusion Criteria:

1. Healthy as judged by a responsible physician with no abnormality identified on a medical evaluation including medical history and physical examination.
2. Males and Females non-smoker aged between 18 years to 60 years.
3. Males and Females weight between 36-75 kilograms.
4. A female is eligible to enter and participate in this study if she is:

   * of non-childbearing potential including pre-menopausal females with documented (medical report verification) hysterectomy or double oophorectomy
   * or postmenopausal defined as 12 months of spontaneous amenorrhea or 6 months of spontaneous amenorrhea with serum follicle stimulating hormone levels >40 milli-International unit (mIU/mL) or 6 weeks postsurgical bilateral oophorectomy with or without hysterectomy
   * or of childbearing potential, has a negative serum pregnancy test at screening and prior to start the study drug in each period, and abstain from sexual intercourse or agrees to using effective contraceptive methods (e.g., intrauterine device, hormonal contraceptive drug, tubal ligation or female barrier method with spermicide) during the study until completion of the follow-up procedures
5. A male is eligible to enter and participate in this study if he: agrees to abstain from (or use a condom during) sexual intercourse with females of childbearing potential or lactating females; or is willing to use a condom/spermicide, during the study until completion of the follow-up procedures.
6. Provide a signed and dated written informed consent prior to study participation.
7. Normal electrocardiogram (ECG) with QTc <450 msec.
8. Willingness and ability to comply with the study protocol for the duration of the trial.

Exclusion Criteria:

1. Females who are pregnant, trying to get pregnant, or are lactating.
2. The subject has evidence of active substance abuse that may compromise safety, pharmacokinetics, or ability to adhere with protocol instructions.
3. A positive pre-study hepatitis B surface antigen, positive hepatitis C antibody, or positive human immunodeficiency virus-1 (HIV-1) antibody result at screening.
4. Subjects with a personal history of cardiac disease, symptomatic or asymptomatic arrhythmias, syncopal episodes, or additional risk factors for torsades de points (heart failure, hypokalemia) or with a family history of sudden cardiac death.
5. A creatinine clearance (CLcr) <70 mL/min as determined by Cockcroft-Gault equation:

   CLcr (mL/min) = (140 - age) * Wt / (72 * Scr) (multiply answer by 0.85 for females) Where age is in years, weight (wt) is in kg, and serum creatinine (Scr) is in units of mg/dL [Cockcroft, 1976].
6. History of alcohol or substance abuse or dependence within 6 months of the study.
7. Use of prescription (especially cytochrome P450 3A4 (CYP3A4) inhibitors or inducers) or non-prescription drugs except paracetamol at doses of up to 2 grams/day, including vitamins (especially vitamin C), herbal and dietary supplements (including St. John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 times the drug half-life (whichever is longer) prior to the first dose of study medication until the completion of the follow-up procedure, unless in the opinion of investigator, the medication will not interfere with the study procedures or compromise subject safety; the investigator will take advice from the manufacturer representative as necessary.
8. The subject has participated in a clinical trial and has received a drug or a new chemical entity within 30 days or 5 half-lives, or twice the duration of the biological effect of any drug (whichever is longer) prior to the first dose of study medication.
9. The subject is unwilling to abstain from ingesting alcohol within 48 hours prior to the first dose of study medication until collection of the final pharmacokinetic sample during each regimen.
10. Subjects who have donated blood to the extent that participation in the study would result in more than 300 mL blood donated within a 30-day period. Plasma donation during the study is not acceptable.
11. Subjects who have a history of allergy to the study drug or drugs of this class, or a history of drug or other allergy that, in the opinion of the investigator, contraindicates participation in the trial. In addition, if heparin is used during pharmacokinetic sampling, subjects with a history of sensitivity to heparin or heparin-induced thrombocytopenia should not be enrolled.
12. Lack of suitability for participation in this study, including but not limited to, unstable medical conditions, systemic disease manifested by tendency to granulocytopenia e.g. rheumatoid arthritis and lupus erythematosus that in the opinion of the investigator would compromise their participation in the trial.
13. Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >1.5 upper limit of normal (ULN)
14. Subjects with history of renal disease, hepatic disease, and/or cholecystectomy
15. Abnormal methaemoglobin level.
16. History of antimalarial drugs use including but not limited to mefloquine, chloroquine, primaquine, artesunate, piperaquine and pyronaridine treatment within 3 months.
17. Subject who received quinacrine in last 30 days.
18. The subject is unwilling to abstain from the consumption of vitamin C 24 hours before and after drug ingestion.
19. History of travel to West or Central Africa, unless it can be verified that subject does not have Loa loa infection.
20. G6PD deficient detected by Beutler's dye test.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2015-10; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events | 1.5 year
  Also including abnormal clinical laboratory, vital signs and corrected QT interval (QTc) prolongation for DHA-PQP

SECONDARY OUTCOMES:
Area under the concentration-time curve AUC(0-∞) | 1.5 year
  Pharmacokinetic parameters
Area under the concentration-time curve AUC(0-last) | 1.5 year
  Pharmacokinetic parameters
Maximal concentration (Cmax) | 1.5 year
  Pharmacokinetic parameters
Elimination clearance (CL/F) | 1.5 year
  Pharmacokinetic parameters
Terminal elimination half-life (t1/2) | 1.5 year
  Pharmacokinetic parameters
Apparent volume of distribution (Vd) for PQ, DHA-PQP, IVM, ABZ. | 1.5 year
  Pharmacokinetic parameters
Pharmacogenetic polymorphisms in case of abnormal drug level | 1.5 year
  Pharmacogenetic polymorphisms in the case of unusually high or low drug levels.
Pharmacokinetic differences of AUC(0-∞) for IVM between venous and capillary blood | 1.5 year
  Pharmacokinetic differences (AUC(0-∞)) for IVM in venous and capillary blood when given alone or together with DHA-PQP.
Pharmacokinetic differences of AUC(0-last) between venous and capillary blood | 1.5 year
  Pharmacokinetic differences (AUC(0-last)) for IVM in venous and capillary blood when given alone or together with DHA-PQP.
Pharmacokinetic differences of Cmax between venous and capillary blood | 1.5 year
  Pharmacokinetic differences (Cmax) for IVM in venous and capillary blood when given alone or together with DHA-PQP.
Mosquito survivorship | 1.5 year
  Duration of survived mosquito post drug drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Dr.Podjanee Jittamala, MD, Principal Investigator — Mahidol University
Locations (1):
- Faculty of Tropical Medicine, Bangkok, Thailand